CLINICAL TRIAL: NCT05413967
Title: Effects of Mills Manipulation Versus NIRSCHL Exercises on Pain, Strength and Function in Patients With Lateral Epicondylitis
Brief Title: Effects of Mills Manipulation and Nirschel Exercises in Patients With Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0129
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis ,Mills Manipulation,NIRSCHL exercises
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mills manipulation in addition to myofasical release therapy (Experimental): mills manipulation
  Interventions: Other: Mills manipulation in addition to myofasical release therapy
- Nirschl exercises in addition to myofascial release therapy (Experimental): Nirschel exercises
  Interventions: Other: Nirschl exercises in addition to myofascial release therapy

INTERVENTIONS:
Other: Mills manipulation in addition to myofasical release therapy — Group A will receive Mills manipulation in addition to myofasical release therapy as baselin
  Arms: Mills manipulation in addition to myofasical release therapy
Other: Nirschl exercises in addition to myofascial release therapy — Group B will receive Nirschl exercises in addition to myofascial release therapy as baseline
  Arms: Nirschl exercises in addition to myofascial release therapy

SUMMARY:
To find effects of mills manipulation versus NIRSCHL EXERCISES on pain ,strength and function in patients with lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis is also known as tennis elbow, an overuse injury that is characterized by pain and tenderness over the lateral epicondyle. The exact etiology has not been well identified, however its commonly associated with repetitive micro trauma from excessive gripping, wrist extension radial deviation or forearm supination. Extensor carpi radialis brevis is the most affected muscle. The aim of this study is to access the effects of mills manipulation versus Nirschl exercises on pain, strength, and function in patients with lateral epicondylitis.

This study will be a Randomized Clinical trial and will be conducted at Pakistan society for rehabilitation of disabled and Mayo Hospital in Lahore. Patients of aged 20-40 years having insidious onset of lateral elbow pain with positive cozens test, Mills test and Maudsley test will be taken. Patients with radial nerve entrapment, cervical radiculopathy and those receiving injections of corticosteroids in last 4 weeks are excluded. The study will include 32 patients randomly divided into two groups A and group B. The study will be completed within the time duration of 10 months after approval of synopsis. Group A will receive mills manipulation while Group B will receive Nirschl exercises. myofascial release therapy will be given to both groups as baseline. both groups will receive 3 sessions per week for 4 weeks (12 sessions), data will be taken by using numeric pain rating scale for pain, hand dynamometer for grip strength and Patient rated tennis elbow evaluation for evaluation of function, at the start of treatment and the end of treatment session. Data will be analysed on SPSS-25.

Key words: lateral epicondylitis, mills manipulation, Nirschl exercises, Patient rated tennis elbow evaluation

ELIGIBILITY:
Inclusion Criteria:

* Pain on lateral epicondyle of humerus when palpated, in the age group of 40-60 years
* Both male and female are included
* Unilateral symptomatic lateral epicondylitis
* Tenderness over palpation of extensor carpi radialis brevis muscle muscle (ECRB)
* Patients with positive cozens test (resisted wrist extension and radial deviation is painful) ,mills test (passive elbow extension & wrist flexion is painful) and maudsley test(resisted middle finger extension is painful)
* Patients having symptoms of lateral epicondylitis for > 3 months

Exclusion Criteria:

* Radial nerve entrapment
* Cervical radiculopathy
* Corticosteroid injection within 4 weeks
* Had received any conservative treatment for lateral epicondylitis in last 4 weeks before entering the study
* Post-surgery patients of lateral epicondylitis
* Radiological findings of extensor tendon calcification

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating scale (NPRS) | 10 months
  The NPRS is used to access the patient intensity of pain. Its score ranges from 0-10 with 0 is being the least painful while 10 is worst. Patient is asked to make three pain ratings, corresponding to current, best and worst pain experienced over the last 24 hours. The average of the 3 ratings is used to represent the patient's level of pain over the previous 24 hours. The NPRS is found to be valid and reliable method for measuring patients perceived pain.
Hand dynamometer | 10 MONTHS
  Hand dynamometer is used to measure the grip strength of the patients. It is considered as a primary clinical measure according to internationally accepted normal hand grip strength ratings in Kgs in patients with various musculoskeletal conditions associated with decreased hand grip strength.
Patient Rated Tennis Elbow Evaluation(PRTEE) | 10 Months
  Patient related tennis elbow evaluation is used to access pain and functional disability of LE patients. The index has two subscales,5 questions are related to pain are scored 0-10, for each question related to pain 0 refereed to no pain while 10 referred as worst pain imaginable. The functional disability scale 0 referred to no difficulty while 10 being referred to unable to do.PRTEE is a valid and reliable instrument for LE patients.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, ppdpt, Principal Investigator — Riphah International University
Locations (1):
- PSRD hospital Ferozpur Road LAHORE, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pitsillides A, Stasinopoulos D. Cyriax Friction Massage-Suggestions for Improvements. Medicina (Kaunas). 2019 May 21;55(5):185. doi: 10.3390/medicina55050185. PMID 31117314
- [Background] Ma KL, Wang HQ. Management of Lateral Epicondylitis: A Narrative Literature Review. Pain Res Manag. 2020 May 5;2020:6965381. doi: 10.1155/2020/6965381. eCollection 2020. PMID 32454922
- [Background] Landesa-Pineiro L, Leiros-Rodriguez R. Physiotherapy treatment of lateral epicondylitis: A systematic review. J Back Musculoskelet Rehabil. 2022;35(3):463-477. doi: 10.3233/BMR-210053. PMID 34397403
- [Background] Yan C, Xiong Y, Chen L, Endo Y, Hu L, Liu M, Liu J, Xue H, Abududilibaier A, Mi B, Liu G. A comparative study of the efficacy of ultrasonics and extracorporeal shock wave in the treatment of tennis elbow: a meta-analysis of randomized controlled trials. J Orthop Surg Res. 2019 Aug 6;14(1):248. doi: 10.1186/s13018-019-1290-y. PMID 31387611